CLINICAL TRIAL: NCT07221266
Title: Changes in Motor Function, Quality of Life, Cardiorespiratory Fitness, and Physiological Markers in People With Parkinson's Disease Following Different Exercise Interventions.
Brief Title: Changes in Movement, Fitness, and Quality of Life in People With Parkinson's Disease After Different Exercise Programs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Katherine Reyes-Brooks, Clinical Assistant Professor, Department of Physical Therapy and Movement Sciences, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2310334
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson's Disease; Exercise intervention; Physical Therapy; Guided Cycling; Non-contact boxing; Aerobic Exercise; Quality of Life; Endothelial Function; Blood Biomarkers; Homocysteine; Vitamin B-12; Inflammation; Oxidative stress; Balance Training; Motor Function
MeSH Terms: conditions — Parkinson Disease; Inflammation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Cycling (Experimental): Participants in this group will complete supervised cycling sessions on a stationary ergometer twice per week for eight weeks. Exercise intensity will be based on each participant's lactate threshold, determined during cardiopulmonary exercise testing (CPET). Each session includes a warm-up, a 40-minute cycling protocol alternating low, moderate, and high intensities, and a cool-down. Heart rate and perceived exertion are continuously monitored.
  Interventions: Behavioral: Guided Cycling
- Non-contact Boxing (Experimental): Participants in this group will take part in a structured non-contact boxing program modeled after the Rock Steady Boxing® framework. Each 60-minute session includes warm-up, agility drills, four rounds of boxing activities (heavy bag, speed bag, mitt work, and double bag), balance circuits, and a cool-down. Sessions are led by a licensed physical therapist and certified boxing coach.
  Interventions: Behavioral: Non-Contact Boxing
- Traditional Physical Therapy (Standard Care) (Active Comparator): Participants in this group will receive standard physical therapy sessions that include aerobic, balance, strengthening, gait, and task-specific training exercises. Each session lasts approximately 60 minutes and is conducted twice weekly for eight weeks under the supervision of a licensed physical therapist. Exercise intensity is set between 60-85% of maximum heart rate, monitored throughout the session.
  Interventions: Behavioral: Traditional Physical Therapy Program (Standard of Care)

INTERVENTIONS:
Behavioral: Guided Cycling — Participants will complete supervised cycling sessions on a stationary ergometer twice per week for eight weeks. Exercise intensity is based on each participant's lactate threshold as determined by cardiopulmonary exercise testing (CPET). Each 60-minute session includes a warm-up, cycling intervals of varying intensity, and a cool-down. Heart rate and perceived exertion are monitored continuously to ensure safety and adherence to prescribed intensity zones.
  Arms: Guided Cycling
Behavioral: Non-Contact Boxing — Non-Contact Boxing Exercise Program
  Participants will engage in a structured, non-contact boxing program modeled after the Rock Steady Boxing® framework. Sessions are held twice weekly for eight weeks and include warm-up activities, agility and coordination drills, four boxing rounds using heavy and speed bags, and a circuit for balance and strength training. Each session concludes with a cool-down. All activities are supervised by licensed physical therapists trained in Parkinson's-specific exercise safety.
  Arms: Non-contact Boxing
Behavioral: Traditional Physical Therapy Program (Standard of Care) — Participants in this group will receive multimodal physical therapy sessions twice per week for eight weeks. Each 60-minute session includes aerobic training (cycling or treadmill), resistance and balance exercises, gait training, and task-specific functional activities such as transfers and turning. Intensity is maintained at 60-85% of maximum heart rate, with continuous heart-rate monitoring. Sessions are led by a licensed physical therapist following standard clinical practice guidelines.
  Arms: Traditional Physical Therapy (Standard Care)

SUMMARY:
Parkinson's disease (PD) is a progressive neurological condition that can affect movement, balance, endurance, and overall quality of life. Exercise is widely recognized as one of the most effective non-pharmacological treatments to help people with PD maintain function and independence. However, not all exercise programs produce the same results, and more research is needed to understand which types of exercise offer the greatest physical and physiological benefits.

This study is designed to examine how different types of structured exercise programs influence motor function, cardiorespiratory fitness, and markers of overall health in individuals with Parkinson's disease. The goal is to better understand how exercise can be used to improve movement, daily activities, and general well-being, as well as how it affects the body at a physiological level.

Participants will be adults diagnosed with idiopathic Parkinson's disease who are medically stable and able to safely participate in exercise. Before beginning the study, participants will complete screening procedures to ensure safety and eligibility. Eligible participants will then be assigned to one of several supervised exercise interventions conducted over a defined period. Each exercise program is designed to improve movement and function but differs in structure or training emphasis (for example, aerobic, functional, or task-specific activity).

Exercise sessions will take place under the supervision of licensed physical therapist. Each session will include warm-up, exercise, and cool-down components. Intensity will be monitored using heart rate and perceived exertion to ensure safety and appropriate challenge. Participants will attend sessions multiple times per week for 8 weeks.

Researchers will collect information about movement abilities, balance, walking, endurance, and daily function using standardized physical therapy assessments such as gait tests, balance measures, and questionnaires related to quality of life at baseline, after 8-weeks of intervention and once more after a 4-week follow-up. In addition, blood samples will be collected to analyze physiological responses to exercise at the same 3 testing intervals. These samples will allow investigators to measure biomarkers related to cardiovascular health, nitric oxide availability, oxidative stress, and inflammation. These biological indicators can help identify how exercise affects underlying health mechanisms that may contribute to improved function in people with Parkinson's disease.

All data will be collected by trained research personnel who are experienced in working with individuals with Parkinson's disease. Participants will be monitored for safety at each session, and any adverse events will be documented and reviewed by the principal investigator and the Institutional Review Board (IRB).

By comparing changes across the different exercise programs, this study aims to determine which interventions have the most meaningful impact on mobility, endurance, and quality of life, as well as which ones produce measurable physiological benefits. Results from this research may help guide physical therapists, rehabilitation professionals, and people with Parkinson's disease in choosing the most effective exercise approaches for maintaining function and promoting overall health.

Ultimately, this project seeks to contribute to the growing evidence that targeted, engaging, and appropriately dosed exercise can play a key role in improving the lives of people living with Parkinson's disease. The findings may also help inform future clinical practice guidelines, community exercise programs, and long-term wellness strategies for individuals with movement disorders.

DETAILED DESCRIPTION:
Background and Rationale Parkinson's disease (PD) is a progressive neurological disorder that affects movement, balance, coordination, and overall function. While medications such as levodopa remain the cornerstone of PD symptom management, they do not slow disease progression or fully address non-motor impairments such as fatigue, autonomic changes, or cardiovascular deconditioning. Exercise has emerged as a powerful, evidence-based intervention that can improve motor performance, cardiovascular function, and quality of life for individuals living with PD. However, the most effective exercise modes and physiological mechanisms underlying these benefits remain unclear.

Previous studies have demonstrated that aerobic training, cycling, and non-contact boxing can enhance mobility and well-being in PD, but few have directly compared these interventions within a single controlled trial. Moreover, little is known about how such exercise programs influence physiological markers of cardiovascular and endothelial health, such as nitric oxide bioavailability, inflammatory cytokines, oxidative stress, and vitamin B-12/homocysteine metabolism. Understanding these effects could provide valuable insight into the systemic adaptations that accompany exercise in PD and help refine individualized therapy prescriptions.

Study Objectives This study aims to compare the effects of three distinct exercise interventions - guided cycling, non-contact boxing, and traditional physical therapy (standard care) - on functional, physiological, and psychosocial outcomes in individuals with Parkinson's disease.

Primary Objectives:

1. To determine which exercise intervention yields the greatest improvements in motor function and balance performance.
2. To assess changes in cardiorespiratory fitness following each intervention.
3. To evaluate improvements in quality of life using validated self-report tools.

   Secondary Objectives:
4. To explore how different exercise types affect physiological markers such as endothelial function (FMD), nitric oxide bioavailability, oxidative stress, inflammatory cytokines (CRP, TNF-α), homocysteine, and vitamin B-12 levels.
5. To assess whether exercise-induced physiological changes are associated with improvements in clinical and functional outcomes.

Study Design

This is a single-site, randomized, controlled, interventional trial conducted in El Paso, Texas, with collaboration between the University of Texas at El Paso (UTEP) and MOVE Therapy Services. Participants will be randomized (computer-generated block randomization) into one of three intervention arms:

1. Guided Cycling Group
2. Non-Contact Boxing Group
3. Traditional Physical Therapy (Standard Care) Group

The total duration for each participant is 15 weeks, consisting of:

* Week 1: Baseline testing
* Weeks 2-9: 8-week intervention (two 60-minute sessions per week)
* Week 10: Post-intervention testing
* Weeks 11-14: Four-week rest/washout
* Week 15: Final follow-up testing

All sessions will be led by licensed physical therapists with assistance from trained Doctor of Physical Therapy (DPT) students. Data collection will occur at UTEP's Rehabilitation Sciences Complex for the cycling and physical therapy groups, and at MOVE Therapy Services for the boxing group.

Intervention Descriptions

1. Non-Contact Boxing:

   This intervention emphasizes large-amplitude, rhythmical, and task-specific movements that combine cognitive, motor, and cardiovascular elements. Sessions include warm-up, boxing rounds (heavy bag, speed bag, mitt work), agility and balance circuits, and cool-down routines. Participants wear gloves, engage in multi-directional footwork, and perform high-intensity drills under therapist supervision. HR and BP are continuously monitored for safety.
2. Guided Cycling:

   This program uses stationary cycle ergometers (Lode Corival) with intensity determined by participants' lactate threshold, established through cardiopulmonary exercise testing (CPET). Each session includes a warm-up, 40-minute cycling component with alternating low, moderate, and high-intensity bouts, and a cool-down. HR and RPE are recorded throughout. Lactate micro-sampling from the earlobe is used periodically to confirm workloads within prescribed zones.
3. Traditional Physical Therapy (Standard Care):

This intervention incorporates multimodal training emphasizing aerobic exercise, resistance and balance training, gait practice, and task-specific functional activities. Intensity is set between 60-85% HRmax, adjusted by perceived exertion and HR monitoring. Each session includes warm-up, treadmill or cycling intervals, balance tasks with and without visual cues, strength training, and community-oriented gait exercises. Safety is ensured through therapist supervision, gait belts, and appropriate rest breaks.

Outcome Measures

Primary Clinical Measures:

* Mini-Balance Evaluation Systems Test (Mini-BESTest)
* 10-Meter Walk Test (10MWT)
* Tinetti Performance-Oriented Mobility Assessment (POMA)
* Parkinson's Disease Questionnaire-39 (PDQ-39)
* Modified Clinical Test of Sensory Interaction in Balance (mCTSIB)

Physiological Outcomes:

* Cardiorespiratory Fitness (VO₂peak)
* Lactate Threshold
* Flow-Mediated Dilation (FMD)
* Blood Biomarkers (NOx, CRP, TNF-α, homocysteine, vitamin B-12, 8-isoprostane)
* Hemodynamic Variables (BP, HR) Sample and Recruitment A total of 45 adults (15 per group) with idiopathic Parkinson's disease, Hoehn and Yahr stages 1-3, and age ≥50 years will be recruited from El Paso and Las Cruces communities through PD support groups, neurologist referrals, flyers, and social media outreach. Inclusion requires independent ambulation and medical clearance for exercise. Exclusion criteria include stroke, myocardial infarction, non-ambulatory status, unmanaged PD medication, or osteoporosis. All participants will provide written informed consent (English or Spanish).

Power analysis using G*Power (Cohen's d = 0.7, α = 0.05, power = 0.8) indicates that 9 participants per group are sufficient; 15 per group will be recruited to account for attrition.

Safety and Risk Management This study is considered minimal risk. All procedures (CPET, venipuncture, boxing, cycling) follow established clinical safety standards. Licensed PTs and CPR/AED-certified personnel will be present at all sessions. Adverse events will be documented and reported to the UTEP IRB. Emergency protocols are in place, and AEDs and communication devices are available within each facility. Participants are instructed to report any discomfort, and sessions will be terminated immediately if needed.

Data Management and Confidentiality All data are coded with unique numeric identifiers. Identifiable information (e.g., consent forms, demographic logs) will be stored separately in a locked cabinet in the PI's office at UTEP. Electronic data will be password-protected and stored on secure UTEP servers. Only the PI will have access to the link between identifiers and coded data. Records will be retained for three years following study completion, then destroyed. No identifiable data will be transmitted outside UTEP.

Statistical Analysis Plan Data will be analyzed using SPSS or equivalent statistical software. Normality will be tested using Shapiro-Wilk. For normally distributed data, two-way repeated-measures ANOVA will be conducted (Group × Time). Non-parametric equivalents (Friedman test) will be applied where assumptions are not met. Post hoc analyses with Bonferroni correction will identify within- and between-group differences. Statistical significance will be set at p < 0.05. Effect sizes will be calculated to quantify magnitude of change.

Expected Significance This research is expected to provide valuable evidence on the comparative effectiveness of three exercise modalities for individuals with Parkinson's disease. By combining clinical, functional, and physiological outcomes, this study will help clarify how different exercise programs influence mobility, cardiovascular health, and biochemical indicators of disease progression.

The findings will directly inform rehabilitation professionals, neurologists, and exercise specialists about the most effective and safe approaches for optimizing health and independence in people with Parkinson's disease. Ultimately, this work may contribute to improved clinical guidelines, personalized exercise prescriptions, and broader access to evidence-based community exercise programs that enhance the lives of people living with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's Disease
2. Independent ambulation
3. Hoehn and Yahr stage of 1-3
4. 50 years of age or older
5. Must speak English or Spanish

Exclusion Criteria:

1. History of stroke
2. History of heart attack
3. Non-ambulatory
4. Hoehn and Yahr of stage 4 or 5
5. Osteoporosis
6. Unmanaged Parkinson's medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-BESTest Total Score | Baseline, Week 10, Week 15.
  The Mini-Balance Evaluation Systems Test (Mini-BESTest) assesses anticipatory control, reactive postural control, sensory orientation, and dynamic gait. Total score range 0-28; higher scores indicate better balance.
Change in VO₂peak (mL/kg/min) During CPET | Baseline, Week 10, Week 15.
  Peak oxygen uptake measured by metabolic cart during graded cycle ergometry; higher values indicate greater cardiorespiratory fitness.
PDQ-39 Summary Index | Baseline, Week 10, Week 15.
  Parkinson's Disease Questionnaire-39 overall summary index; lower scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
10-Meter Walk Test (10MWT) Speed | Baseline, Week 10, Week 15.
  The 10MWT measures gait speed in meters per second over a 10-meter distance. Increased speed indicates improved walking ability.
Tinetti Performance-Oriented Mobility Assessment (POMA) Score | Baseline, Week 10, Week 15.
  The POMA evaluates balance and gait function. Scores range from 0-28, with higher scores reflecting improved mobility and reduced fall risk.
Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) Score | Baseline, Week 10, Week 15.
  The mCTSIB assesses postural stability under four sensory conditions. Longer hold times indicate improved sensory integration and balance.
Flow-Mediated Dilation (FMD) Percentage | Baseline, Week 10, Week 15.
  Endothelial function will be evaluated by ultrasound measurement of brachial artery diameter changes after occlusion. Greater FMD percentage indicates improved vascular function.
Blood Biomarker Levels (NOx, CRP, TNF-α, Homocysteine, Vitamin B-12, 8-Isoprostane) | Baseline, Week 10, Week 15.
  Venous blood samples will be analyzed for nitric oxide bioavailability (NOx), C-reactive protein (CRP), tumor necrosis factor-alpha (TNF-α), homocysteine, vitamin B-12, and oxidative stress marker 8-isoprostane. These biomarkers reflect inflammatory and metabolic responses to exercise.
Blood Lactate Concentration During CPET | Baseline, Week 10, Week 15.
  Blood lactate levels (mmol/L) will be collected through micro-sampling from the earlobe during graded exercise testing. A rightward shift in lactate threshold indicates improved metabolic efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Reyes-Brooks, PT, DPT, Principal Investigator — University of Texas, El Paso
Locations (2):
- United States (2):
  - University of Texas at El Paso Doctor of Physical Therapy and Movement Sciences Building, El Paso, Texas
  - Move Therapy Services, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available without identifiers upon request.

REFERENCES:
- [Background] Larson D, Yeh C, Rafferty M, Bega D. High satisfaction and improved quality of life with Rock Steady Boxing in Parkinson's disease: results of a large-scale survey. Disabil Rehabil. 2022 Oct;44(20):6034-6041. doi: 10.1080/09638288.2021.1963854. Epub 2021 Sep 9. PMID 34498995
- [Background] Gurovich AN, Avery JC, Holtgrieve NB, Braith RW. Flow-mediated dilation is associated with endothelial oxidative stress in human venous endothelial cells. Vasc Med. 2014 Aug;19(4):251-256. doi: 10.1177/1358863X14537546. Epub 2014 Jun 10. PMID 24916471
- [Background] Amara AW, Memon AA. Effects of Exercise on Non-motor Symptoms in Parkinson's Disease. Clin Ther. 2018 Jan;40(1):8-15. doi: 10.1016/j.clinthera.2017.11.004. Epub 2017 Dec 1. PMID 29198450
- [Background] Sangarapillai K, Norman BM, Almeida QJ. Boxing vs Sensory Exercise for Parkinson's Disease: A Double-Blinded Randomized Controlled Trial. Neurorehabil Neural Repair. 2021 Sep;35(9):769-777. doi: 10.1177/15459683211023197. Epub 2021 Jun 13. PMID 34121511
- [Background] Fang YC, Hsieh YC, Hu CJ, Tu YK. Endothelial Dysfunction in Neurodegenerative Diseases. Int J Mol Sci. 2023 Feb 2;24(3):2909. doi: 10.3390/ijms24032909. PMID 36769234
- [Background] Adams JD Jr, Odunze IN. Oxygen free radicals and Parkinson's disease. Free Radic Biol Med. 1991;10(2):161-9. doi: 10.1016/0891-5849(91)90009-r. PMID 2016074
- [Background] Osborne JA, Botkin R, Colon-Semenza C, DeAngelis TR, Gallardo OG, Kosakowski H, Martello J, Pradhan S, Rafferty M, Readinger JL, Whitt AL, Ellis TD. Physical Therapist Management of Parkinson Disease: A Clinical Practice Guideline From the American Physical Therapy Association. Phys Ther. 2022 Apr 1;102(4):pzab302. doi: 10.1093/ptj/pzab302. PMID 34963139
- [Background] Ridgel AL, Vitek JL, Alberts JL. Forced, not voluntary, exercise improves motor function in Parkinson's disease patients. Neurorehabil Neural Repair. 2009 Jul-Aug;23(6):600-8. doi: 10.1177/1545968308328726. Epub 2009 Jan 8. PMID 19131578
- [Background] Osborne JA, Botkin R, Colon-Semenza C, DeAngelis TR, Gallardo OG, Kosakowski H, Martello J, Pradhan S, Rafferty M, Readinger JL, Whitt AL, Ellis TD. Correction to: Osborne JA, Botkin R, Colon-Semenza C, et al. Physical Therapist Management of Parkinson Disease: A Clinical Practice Guideline From the American Physical Therapy Association. Phys Ther. 2022;102:pzab302. https://doi.org/10.1093/ptj/pzab302. Phys Ther. 2022 Aug 1;102(8):pzac098. doi: 10.1093/ptj/pzac098. No abstract available. PMID 36029042